CLINICAL TRIAL: NCT05923060
Title: Noninvasive Imaging Techniques to Monitor Photosensitizer and Singlet Oxygen Levels During Photodynamic Therapy of Actinic Keratoses
Brief Title: Imaging Techniques to Monitor Photosensitizer and sO2 Levels During Photodynamic Therapy of Actinic Keratoses
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CASE6622; R44CA250727 (NIH)
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Actinic Keratoses
Keywords: Actinic Keratoses; Red Light; Photodynamic Therapy; Protoporphyrin IX
MeSH Terms: conditions — Keratosis, Actinic | interventions — Aminolevulinic Acid; Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Standard PDT + topical aminolevulinate + red light illumination (Experimental): Standard PDT using topical aminolevulinate followed by red light illumination for actinic keratosis. A region of interest (ROI) on the skin of the arms, hands, legs, or feet will be selected for monitoring. This ROI will be marked and baseline measurements will be taken. The topical drug Levulan (ALA) will be applied to the ROI and other areas being treated, and covered with plastic wrap. Prior to red light illumination, post topical measurements and baseline values will be performed to measure PpIX and sO2. Red light illumination will follow, and sO2 phosphorescence will be recorded continuously from the ROI. After, a post-PpIX measurement will be taken.
  Interventions: Drug: Topical Aminolevulinate; Procedure: Photodynamic therapy (PDT); Procedure: Red light illumination

INTERVENTIONS:
Drug: Topical Aminolevulinate — Topical Levulan Kerastick is applied to actinic keratoses.
  Other Names: Levulan Kerastick; Aminolevulinic Acid; Levulan
Procedure: Photodynamic therapy (PDT) — PDT is a technique that combines a photosensitizing drug and an intense light source to kill tumor cells.
Procedure: Red light illumination — To occur post-PTD; used for activation of ALA during photodynamic therapy.

SUMMARY:
The purpose of the study is to test a new video device for actinic keratoses. The device takes images of your skin lesions during the treatment, to learn whether this device can predict how well the treatment is working.

DETAILED DESCRIPTION:
This intervention is designed to help establish what the optimal conditions are for treating actinic keratoses with photodynamic therapy (PDT). The primary outcome of this study is to determine whether the rate of singlet oxygen (sO2) production and/or the initial intralesional photosensitize (PpIX) levels, can predict the clinical responsiveness of AK lesions to PDT. Participants will receive standard red light PDT treatment, except that lesions will be carefully counted beforehand. During the window of red light illumination, photos and a video of one area of skin will be taken to allow us to monitor the progress of the treatment. Any remaining lesions will be counted upon follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have at least 10 Actinic Keratoses lesions on the arms of legs, and with two AK lesions close enough to be seen together within a selected region of interest (ROI)
* Participants must be able to understand and are willing to sign a written informed consent document

Exclusion Criteria:

* Female participants cannot be or become pregnant, nor can be nursing while on this study
* Using any topical treatment on their AKs; must stop at least one month prior
* Currently undergoing treatment for other cancers with medical or radiation therapy
* Patients with a known hypersensitivity to 5-aminolevulinic acid or any component of the study material
* Patients with history of a photosensitivity disease, such as porphyria cutanea tarda

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-25 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Lesion Clearance | 3 months post PDT treatment.
  Based on the rate of sO2 production, and/or the initial level of PpIX, is significantly correlated with the clinical responsiveness of AK lesions to PDT treatment. The clinical responsiveness will be measured by the decrease in the number of lesions
Noninvasive optical measurements of photosensitizer (PpIX) in lesions | 3 months post PDT treatment.
  To determine whether the initial level of PpIX can predict the clinical responsiveness of AK lesions to PDT treatment. The clinical responsiveness will be measured by the change in PpIX value before and after red light illumination.
Noninvasive optical measurements of singlet oxygen (sO2) in lesions. | 3 months post PDT treatment.
  To determine whether the rate of sO2 production can predict the clinical responsiveness of AK lesions to PDT treatment. The clinical responsiveness will be measured by the change in sO2 value before and after red light illumination.

SECONDARY OUTCOMES:
Noninvasive optical measurements variability of photosensitizer (PpIX) in lesions | 3 months post PDT treatment.
  To characterize the variability in PpIX production between similarly-sized lesions. This will be measured by the accumulation of PpIX.
Noninvasive optical measurements variability of singlet oxygen (sO2) in lesions | 3 months post PDT treatment.
  To characterize the variability in sO2 generation between similarly-sized lesions, and to test whether production of sO2 during PDT correlates with the amount of photosensitizer available in AK lesions. This will be measured by sO2 production, measured in real-time by sO2 dosimeter.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Maytin, MD, PhD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in publication
Supporting Information: Analytic Code
Access Criteria: Cleveland Clinic will share de-identified optical digital code from the fluorescence instrument with Physical Sciences, Inc where it will be processed for final spectral analysis